CLINICAL TRIAL: NCT04443231
Title: Prospective Clinical Study of Retinal Microvascular Alteration After ICL Implantation
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: tch0101
Record Dates: First submitted 2020-03-17; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2019-07

CONDITIONS: Adolescent; Adult; Human; Male; Female; Follow-up Studies; Prospective Studies; Lens Implantation, Intraocular; Myopia; Phakic Intraocular Lenses; Retinal Vessels; Postoperative Period; Preoperative Period; Tomography, Optical Coherence
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Optical Coherence Tomography Angiography — AngioVue (Optovue, Fremont, CA, USA) was used to capture the OCTA images before ICL surgery and at 3 months follow-up.

SUMMARY:
To observe the retinal microvascular alteration during 3 months follow-up after Implantable Collamer Lens (ICL) operation in moderate and high myopia patients using quantitative optical coherence tomography angiography (OCTA) analysis.

DETAILED DESCRIPTION:
The study object is moderate and high myopia patients, underwent ICL implantation. OCTA was used to image the superficial and deep retinal vascular plexuses before ICL implantation surgery and at 3 months follow-up. OCTA images were corrected for magnification, skeletonized, separated the large vessels and partitioned. Retinal microvascular density was measured by using fractal dimension analysis. The aim of this study was to uncover potential retinal vascular network alterations induced by ICL implantation surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years old;
* Binocular myopia, with a refraction of greater than -3 diopters (D);
* anterior chamber depth (ACD, measured from the endothelium to the crystalline lens) > 2.8 mm;
* corneal endothelial cell count (cECC) ≥ 2000 cells/mm2;
* stable refraction at least 1 year before surgery;
* unsatisfactory vision with contact lenses or spectacles.

Exclusion Criteria:

* history of intraocular surgery
* other ocular pathology (uveitis, glaucoma, cataract, keratoconus, severe dry eye, etc.)
* other serious systemic disease (diabetes, uncontrolled hypertension, severe hyperthyroidism, etc.).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Moderate and high myopia patients, underwent ICL implantation surgery at the Department of Ophthalmology, Peking University Third Hospital
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Retinal microvessels density | 3 months postoperatively
  Retinal microvessels density was measured with fractal dimension analysis by using Matalb (The Mathworks, Inc., Natick, MA, USA)

SECONDARY OUTCOMES:
Best corrected visual acuity | 3 months postoperatively
  BCVA was evaluated by decimal Snellen and converted to the logarithm of the minimum angle of resolution (logMAR) for statistical analysis.
Mean refractive spherical equivalent | 3 months postoperatively
  MRSE = Spherical power + 0.5 * Cylindrical power
Intraocular pressure | 3 months postoperatively
  The IOP was measured using a non-contact tonometer (CT-80; Topcon, Tokyo, Japan).
Vault | 3 months postoperatively
  The central vault of the ICL (distance from posterior surface of ICL to the crystalline lens) was measured using Optical Coherence Tomography (Visante; Carl Zeiss Meditec, Jena, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, PhD, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanders DR, Doney K, Poco M; ICL in Treatment of Myopia Study Group. United States Food and Drug Administration clinical trial of the Implantable Collamer Lens (ICL) for moderate to high myopia: three-year follow-up. Ophthalmology. 2004 Sep;111(9):1683-92. doi: 10.1016/j.ophtha.2004.03.026. PMID 15350323
- [Result] Yang Y, Wang J, Jiang H, Yang X, Feng L, Hu L, Wang L, Lu F, Shen M. Retinal Microvasculature Alteration in High Myopia. Invest Ophthalmol Vis Sci. 2016 Nov 1;57(14):6020-6030. doi: 10.1167/iovs.16-19542. PMID 27820633
- [Result] Li M, Yang Y, Jiang H, Gregori G, Roisman L, Zheng F, Ke B, Qu D, Wang J. Retinal Microvascular Network and Microcirculation Assessments in High Myopia. Am J Ophthalmol. 2017 Feb;174:56-67. doi: 10.1016/j.ajo.2016.10.018. Epub 2016 Nov 4. PMID 27818204